CLINICAL TRIAL: NCT05222191
Title: Spironolactone in Chronic Kidney Disease Enabled by Chlorthalidone: A Pilot Randomized Control Trial
Brief Title: Spironolactone in CKD Enabled by Chlorthalidone: PILOT
Acronym: SPICE PILOT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indiana Institute for Medical Research (Other)
Responsible Party: Principal Investigator, Rajiv Agarwal, Principal Investigator, Indiana Institute for Medical Research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12672
Record Dates: First submitted 2022-01-18; First posted 2022-02-03 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Renal Insufficiency; Chronic Hypertension
Keywords: Spironolactone; Chlorthalidone; Chronic Kidney Disease; Hypertension; Thiazide Diuretic; Potassium Sparring Diuretic
MeSH Terms: conditions — Renal Insufficiency; Renal Insufficiency, Chronic; Hypertension | interventions — Spironolactone; Chlorthalidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spironolactone + Placebo (Active Comparator): Subjects with stage 3B/4 chronic kidney disease and poorly controlled hypertension will be randomized into two groups: one receiving spironolactone and placebo and one receiving spironolactone and chlorthalidone. At randomization, subjects will begin at 25 mg spironolactone and 6.25 mg placebo/chlorthalidone daily.
  Interventions: Drug: Spironolactone; Drug: Placebo
- Spironolactone + Chlorthalidone (Experimental): Subjects with stage 3B/4 chronic kidney disease and poorly controlled hypertension will be randomized into two groups: one receiving spironolactone and placebo and one receiving spironolactone and chlorthalidone. At randomization, subjects will begin at 25 mg spironolactone and 6.25 mg placebo/chlorthalidone daily.
  Interventions: Drug: Spironolactone; Drug: Chlorthalidone

INTERVENTIONS:
Drug: Spironolactone — Study drugs will be increased if goal blood pressure is not achieved and/or serum potassium is not in safe clinical range (dosage of chlorthalidone/placebo not to exceed 25 mg daily; dosage of spironolactone not to exceed 50 mg daily).
Drug: Chlorthalidone — Study drugs will be increased if goal blood pressure is not achieved and/or serum potassium is not in safe clinical range (dosage of chlorthalidone/placebo not to exceed 25 mg daily; dosage of spironolactone not to exceed 50 mg daily).
  Arms: Spironolactone + Chlorthalidone
Drug: Placebo — Study drugs will be increased if goal blood pressure is not achieved and/or serum potassium is not in safe clinical range (dosage of chlorthalidone/placebo not to exceed 25 mg daily; dosage of spironolactone not to exceed 50 mg daily).
  Arms: Spironolactone + Placebo

SUMMARY:
Highly prevalent among patients with chronic kidney disease (CKD) and poorly controlled blood pressure (BP), is a modifiable risk factor to abrogate both kidney failure progression and cardiovascular (CV) disease. Spironolactone (SPL), a mineralocorticoid receptor antagonist, is widely used to treat resistant hypertension, however one of the most common side effects is an increase of serum potassium (K). This side effect occurs frequently in those who suffer from CKD. Alternatively, chlorthalidone (CTD) is a thiazide-like diuretic used for treating hypertension and decreases serum K. In this pilot study, our goal is to assess whether the combination of SPL and CTD can improve BP control, while also reducing the risk of hyperkalemia over a period of 12 weeks. We hypothesize that among patients with CKD and poorly controlled hypertension, compared to SPL and placebo, treatment over 12 weeks with CTD will counter the hyperkalemia effect of SPL, and therefore the combination of SPL with CTD will result in a lower BP. This pilot study will be performed at Richard L. Roudebush VA in Indianapolis, Indiana.

DETAILED DESCRIPTION:
This is a placebo-controlled, double-blind, randomized controlled trial of spironolactone (SPL) and chlorthalidone (CTD) in patients with CKD and poorly controlled hypertension

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years.
2. GFR estimated by CKD-EPI formula < 45 ml/min/1.73 m2 but ≥ 15 mL/min/1.73 m2 using IDMS-calibrated creatinine.
3. Hypertension. Using AOBP monitoring, BP of ≥ 130/80 mmHg.
4. Treatment with antihypertensive drugs: This would require the use of at least one antihypertensive drug. One of the drugs should be either an ACE inhibitor or ARB or a beta-blocker at the time of randomization.
5. Serum K 3.5 to 5.2 mEq/L at the time of randomization. In patients with eGFR < 45 ml/min/1.73 m2 and serum K > 5.2 mEq/L

Exclusion Criteria:

1. Use of spironolactone, eplerenone, amiloride, triamterene, thiazides, or thiazide-like drugs or the use of K supplements or K binders in the previous 12 weeks.
2. Expected to receive renal replacement therapy within the next 6 months.
3. Myocardial infarction, heart failure hospitalization, or stroke ≤ 12 weeks prior to randomization.
4. Pregnant or breastfeeding women or women who are planning to become pregnant or those not using a reliable form of contraception (oral contraceptives. condoms and diaphragms will be considered reliable).
5. Known hypersensitivity to thiazide or spironolactone.
6. Clinic AOBP <110 mmHg systolic at their first visit

Ages: 19 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-12-12 (Estimated); Study Completion 2023-12-12 (Estimated)

PRIMARY OUTCOMES:
Change in Systolic Automated Office Blood Pressure from baseline to 12 weeks between arms | Baseline to 12 Weeks

SECONDARY OUTCOMES:
Change in logarithmically transformed albumin/creatinine ratio from baseline to 12 weeks between arms | Baseline to 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Agarwal, MD, Principal Investigator — Indiana Institute for Medical Research; Roudebush VA Medical Center
Locations (1):
- Richard L Roudebush VA Medical Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No